CLINICAL TRIAL: NCT06674759
Title: Efficacy and Safety of Tongren-Dahuoluo Bolus in Patients with Knee Osteoarthritis: a Randomized, Double-blind, Placebo-controlled Clinical Study
Brief Title: Efficacy and Safety of Tongren-Dahuoluo Bolus in Patients with Knee Osteoarthritis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Quan Jiang, Director，Devision of Rheumatology, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-170-YW-01
Record Dates: First submitted 2024-10-30; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Knee Osteoarthritis (Knee OA)
Keywords: Tongren-Dahuoluo Bolus; Knee osteoarthritis (Knee OA)
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment of Tongren Dahuoluo Pills (Experimental)
  Interventions: Drug: Tongren-Dahuoluo Bolus
- Treatment of Tongren-Dahuoluo Bolus Placebo (Placebo Comparator)
  Interventions: Drug: Tongren-Dahuoluo Bolus Placebo

INTERVENTIONS:
Drug: Tongren-Dahuoluo Bolus — 0.72g,2 times a day, oral, for 24 weeks.
  Arms: Treatment of Tongren Dahuoluo Pills
Drug: Tongren-Dahuoluo Bolus Placebo — 0.72g,2 times a day, oral, for 12 weeks.
  Arms: Treatment of Tongren-Dahuoluo Bolus Placebo

SUMMARY:
The clinical trial has a research cycle of 24 weeks. The first 12 weeks are multicenter, randomized, double-blind, controlled trials. A total of 72 patients with knee osteoarthritis with liver-kidney deficiency syndrome and/or cold-dampness arthralgia syndrome are planned to be enrolled and randomly assigned to the control group (Tongren-Dahuoluo Bolus) and the treatment group (Tongren-Dahuoluo Bolus Placebo) in a 1:1 ratio. The purpose is to compare the safety and efficacy of Tongren-Dahuoluo Bolus and placebo in treating knee osteoarthritis. A long-term blind extension study will be conducted in the next 12 weeks. All subjects will take Tongren-Dahuoluo Bolus orally to evaluate the long-term safety, tolerability, and efficacy of Tongren-Dahuoluo Pills in treating patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 40 to 75 years old;
2. Meet the diagnostic criteria for primary knee osteoarthritis (KOA) (the diagnostic criteria refer to the 1995 American College of Rheumatology classification criteria for knee osteoarthritis);
3. Meet the diagnostic criteria for liver and kidney deficiency and (or) cold and dampness obstruction in the group standard of the Chinese Association of Traditional Chinese Medicine "Guidelines for Combination of Osteoarthritis Symptoms";
4. X-ray examination of the joints is graded as I to III (knee joint Kellgren/Lawrence e scoring standard);
5. Knee pain score ≥40mm in the past week (assessed by VAS standard);

Exclusion Criteria:

1. Patients with other rheumatic diseases such as Sjögren's syndrome, gout, rheumatoid arthritis, or a history of human immunodeficiency virus (HIV);
2. Patients with severe lesions of important organs such as the heart, liver, and kidney, abnormal liver function (alanine or aspartate aminotransferase or glutamine transpeptidase>1.5 times the upper limit of normal value); or abnormal renal function (serum creatinine level> upper limit of normal value); white blood cell (white blood cell, WBC) or platelet (platelet, PLT) below the lower limit of normal value; or diabetic patients with poor blood sugar control in the recent period (glycosylated hemoglobin>8.0%);
3. Patients with suppurative, nonspecific, and other infectious knee arthritis;
4. Patients with traumatic, villonodular pigmentation and other lesions with knee synovium as the main lesions;
5. Patients with advanced joint deformity or disability; A randomized controlled study on Tongren Dahuoluowan in the treatment of knee osteoarthritis Version number: 2023009P8A01 Version date: December 23, 2022
6. Allergic constitution and allergic to the test drug;
7. Pregnant, pregnant, or lactating women;
8. Those who are taking antidepressants, anticonvulsants, opioids, sedatives and glucocorticoids;
9. Patients who have received intra-articular treatment with sodium hyaluronate within 4 weeks before screening; those who have taken drugs containing chondroitin sulfate/glucosamine/diacerein within 3 months before screening; those who have used biological agents within 3 months before screening;
10. Patients with organ failure symptoms;
11. Those who have participated in any other drug trials within 1 month before selection;
12. Those who the researcher believes are not eligible to join this clinical trial

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-01-10 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes from Baseline to week 24 in Visual Analog Scale (VAS)score | 0 week, 4 weeks,12 weeks, 24 weeks
  VAS scores ranges from 0 to 100, with higher scores indicating heavier pain

SECONDARY OUTCOMES:
Changes in the 30s-CST frequency (30-second chair sit-stand test) of the experimental group relative to the baseline and control group at the 4th, 12th, and 24th weeks; | 0 week, 4 weeks,12 weeks, 24 weeks
Changes in knee osteoarthritis index (WOMAC score) at week 4, week 12, and week 24 relative to baseline and control group | 0 week, 4 weeks,12 weeks, 24 weeks
Changes in TCM syndrome score evaluation at week 4, week 12, and week 24 relative to baseline and control group; | 0 week, 4 weeks,12 weeks, 24 weeks
Changes in KOOS scores of knee injury and osteoarthritis outcomes at weeks 4, 12, and 24 relative to baseline and the control group | 0 week, 4 weeks,12 weeks, 24 weeks
Changes in SF-12 at week 4, week 12, and week 24 relative to baseline and control group | 0 week, 4 weeks,12 weeks, 24 weeks
Changes in serum inflammatory indicators (CRP) relative to baseline and control group at week 4, week 12, and week 24 | 0 week, 4 weeks,12 weeks, 24 weeks
  CRP in μg/L
Changes in serum inflammatory indicators (ESR) relative to baseline and control group at week 4, week 12, and week 24 | 0 weeks, 4 weeks,12 weeks, 24 weeks
  ESR in mm/h
MRI examination of the knee joint (target joint) at the time of enrollment and at week 24 to examine the changes in bone marrow edema, joint effusion, synovitis, cartilage volume and composition relative to the baseline and control group | 0 week, 4 weeks,12 weeks, 24 weeks

IPD SHARING:
Plan to Share IPD: No
Ethical Considerations: Adhering to ethical guidelines that prioritize patient consent and data protection.
  Lack of Consent: Patients may not have consented to share their data publicly.